CLINICAL TRIAL: NCT02433483
Title: A Phase II Study of Microtransplantation in Patients With Refractory or Relapsed Hematologic Malignancies
Brief Title: Microtransplantation to Treat Refractory or Relapsed Hematologic Malignancies in Younger Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed due to poor accrual and because of competing protocols.
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Cookies for Kids' Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITREL; NCI-2015-00691 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-04-29; First posted 2015-05-05 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: Adolescent; Children; Microtransplant; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Cytarabine; Methotrexate; Fecal Microbiota Transplantation; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Myeloid Malignancies (Experimental): Includes participants with AML and MDS. Participants receive chemotherapy based on diagnosis followed by infusion of donor HPC-A.
  Participants with CNS disease receive weekly age-adjusted intrathecal triples therapy until the cerebrospinal fluid becomes free of leukemia (minimum of 4 doses).
  Interventions:
  * Cycle 1: cytarabine, HPC-A donor infusion
  * Cycle 2: Participants who have at least a partial response to Cycle 1 are eligible to receive Cycle 2: cytarabine, HPC-A infusion
  Interventions: Drug: Cytarabine; Drug: Intrathecal Triples; Biological: HPC-A

INTERVENTIONS:
Drug: Cytarabine — Given by either intrathecal (IT) or intravenous (IV) route.
  Other Names: Cytosine arabinoside; Ara-C; Cytosar®
Drug: Intrathecal Triples — given IT.
  Other Names: ITMHA; Methotrexate/hydrocortisone/cytarabine
Biological: HPC-A — Given IV.
  Other Names: Donor infusion; Hematopoietic Progenitor Cell, Apheresis

SUMMARY:
Allogeneic transplant can sometimes be an effective treatment for leukemia. In a traditional allogeneic transplant, patients receive very high doses of chemotherapy and/or radiation therapy, followed by an infusion of their donor's bone marrow or blood stem cells. The high-dose chemotherapy drugs and radiation are given to remove the leukemia cells in the body. The infusion of the donor's bone marrow or blood stem cells is given to replace the diseased bone marrow destroyed by the chemotherapy and/or radiation therapy. However, there are risks associated with allogeneic transplant. Many people have life-threatening or even fatal complications, like severe infections and a condition called graft-versus-host disease, which is caused when cells from the donor attack the normal tissue of the transplant patient.

Recently, several hospitals around the world have been using a different type of allogeneic transplant called a microtransplant. In this type of transplant, the donor is usually a family member who is not an exact match. In a microtransplant, leukemia patients get lower doses of chemotherapy than are used in traditional allogeneic transplants. The chemotherapy is followed by an infusion of their donor's peripheral blood stem cells. The objective of the microtransplant is to suppress the bone marrow by giving just enough chemotherapy to allow the donor cells to temporarily engraft (implant), but only at very low levels. The hope is that the donor cells will cause the body to mount an immunologic attack against the leukemia, generating a response called the "graft-versus-leukemia" effect or "graft-versus-cancer" effect, without causing the potentially serious complication of graft-versus-host disease.

With this research study, the investigators hope to find out whether or not microtransplantation will be a safe and effective treatment for children, adolescents and young adults with relapsed or refractory hematologic malignancies

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To assess the safety and feasibility of standard chemotherapy plus GCSF-mobilized Hematopoietic Progenitor Cell, Apheresis (HPC-A) in pediatric patients with relapsed or refractory hematologic malignancies.
* To estimate the response rates to standard chemotherapy plus GCSF-mobilized HPC-A in pediatric patients with relapsed or refractory hematologic malignancies.

SECONDARY OBJECTIVES:

* To describe the event-free and overall survival of patients treated with standard chemotherapy plus GCSF-mobilized HPC-A.
* To estimate the time to neutrophil and platelet recovery after treatment with standard chemotherapy plus GCSF-mobilized HPC-A.
* To determine the cumulative incidence of acute and chronic graft-versus-host disease (GVHD).

OTHER PRESPECIFIED OBJECTIVES:

* To characterize donor chimerism and microchimerism.

Patients will receive standard chemotherapy followed by infusion of donor peripheral blood mononuclear cells 2 days after the completion of chemotherapy. Patients who have at least a partial response are eligible to receive a second cycle.

Diagnostic lumbar puncture and intrathecal (IT) chemotherapy will be given prior to cycle 1. Patients without evidence of central nervous system (CNS) leukemia will receive no further IT therapy during cycle 1. Patients with CNS disease will receive weekly IT therapy (age-adjusted methotrexate, hydrocortisone, and cytarabine) until the cerebrospinal fluid (CSF) becomes free of leukemia (minimum of 4 doses).

Bone marrow aspiration (BMA) and biopsy to assess response will be performed on approximately day 29 of therapy.

For hematopoietic stem cell mobilization, donors will receive G-CSF (Filgrastim) (Neupogen®) each day for 5 days given subcutaneously (SQ) prior to HPC-A collected by leukapheresis on day 6.

ELIGIBILITY:
INCLUSION CRITERIA - AML and MDS PARTICIPANTS

* Participants must have a diagnosis of AML or myelodysplastic syndrome (MDS), ALL, and must have disease that has relapsed or is refractory to chemotherapy, or that has relapsed after HSCT.

  * Refractory disease is defined as persistent disease after at least two courses of induction chemotherapy.
  * Patients with AML must have ≥ 5% leukemic blasts in the bone marrow or have converted from negative minimal residual disease (MRD) status to positive MRD status in the bone marrow as assessed by flow cytometry. If an adequate bone marrow sample cannot be obtained, patients may be enrolled if there is unequivocal evidence of leukemia in the peripheral blood.
* Participant is ≤ 21 years of age (i.e., has not reached 22nd birthday).
* Adequate organ function defined as the following:

  * Total bilirubin ≤ upper limit of normal (ULN) for age, or if total bilirubin is > ULN, direct bilirubin is ≤ 1.5 mg/dL
  * AST (SGOT)/ALT (SGPT) < 5 x ULN
  * Calculated creatinine clearance > 50 ml/min/1.73m^2 as calculated by the Schwartz formula for estimated glomerular filtration rate >
  * Left ventricular ejection fraction ≥ 40% or shortening fraction ≥ 25%.
* Has an available HPC-A donor.
* Performance status: Lansky ≥ 50 for patients who are ≤ 16 years old and Karnofsky ≥ 50% for patients who are > 16 years old.
* Does not have an uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines is acceptable.
* Patient has fully recovered from the acute effects of all prior therapy and must meet the following criteria.

  * At least 14 days must have elapsed since the completion of myelosuppressive therapy.
  * At least 24 hours must have elapsed since the completion of hydroxyurea, low-dose cytarabine (up to 200 mg/m^2/day), and intrathecal chemotherapy.
  * At least 30 days must have elapsed since the use of investigational agents.
  * For patients who have received prior HSCT, there can be no evidence of GVHD and greater than 60 days must have elapsed since the HSCT. Patients cannot be receiving therapy, including steroids, for GVHD.
* Post-menarchal female has had negative serum pregnancy test within 7 days prior to enrollment.
* Male or female of reproductive potential has agreed to use effective contraception for the duration of study participation.
* Not breastfeeding

INCLUSION CRITERIA - HPC-A CELL DONOR

* At least 18 years of age.
* Family member (first degree relatives).
* Not pregnant as confirmed by negative serum or urine pregnancy test within 7 days prior to enrollment (if female).
* Not breast feeding.
* Meets donation eligibility requirements as outlined by 21 CFR 1271.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E. Rubnitz, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two participants and 2 bone marrow or blood stem cell donors were enrolled at St. Jude Children's Research Hospital between May 2015 and July 2015. The donors do not undergo protocol therapy interventions and are not included in the results reporting provided here.
Groups:
- Myeloid Malignancies: Includes participants with AML and MDS. Participants receive chemotherapy based on diagnosis followed by infusion of donor HPC-A.
  Participants with CNS disease receive weekly age-adjusted intrathecal triples therapy until the cerebrospinal fluid becomes free of leukemia (minimum of 4 doses).
  Interventions:
  * Cycle 1: cytarabine, HPC-A donor infusion
  * Cycle 2: Participants who have at least a partial response to Cycle 1 are eligible to receive Cycle 2: cytarabine, HPC-A infusion
  Cytarabine: Given by either intrathecal (IT) or intravenous (IV) route.
  Intrathecal Triples: given IT.
  HPC-A: Given IV.
Period: Overall Study
Arm/Group | Myeloid Malignancies
Started | 2
Completed | 0
Not Completed | 2
Not completed — Unacceptable toxicity | 1
Not completed — Other antineoplastic therapy/HSCT | 1

BASELINE CHARACTERISTICS:
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 7.45 [2.66 to 12.29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by Stratum Who Complete 2 Cycles of Therapy
Description: If two or more patients die from causes other than leukemia progression or experience ≥ Grade 3 GVHD that is associated with detectable donor chimerism due to this protocol, or demonstrate persistent engraftment defined as >5% donor chimerism at the time of count recovery (ANC > 0.3 x 10^9/L and platelet count > 30 x 10^/L), then the cohort will close due to intolerability. Any subject who transfers to transplant prior to completion of two courses without experiencing an unacceptable toxicity is considered inevaluable for purposes of evaluating tolerability. Accrual will be halted for intolerability if there are two or more failures in tolerability among the first six subjects who are evaluable for tolerability.
Time Frame: At the end of therapy cycle 2 (approximately 2-3 months)
Measure: Count of Participants; unit: Participants
Groups:
- Myeloid Malignancies: Includes participants with AML and MDS. Participants receive chemotherapy based on diagnosis followed by infusion of donor HPC-A.
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Proportion of Participants Who Experience Therapeutic Success
Description: All patients will be counted towards this two-stage design. Therapeutic success for patients at time of enrollment is defined as:
  * Patients with fewer than 5% blasts, a ≥ 10-fold decrease in level of minimal residual disease after completion of 1 or 2 cycles of therapy.
  * Patients with greater than 5% in leukemic blasts in the marrow, achieving CR or CRi after completion of 1 or 2 cycles of therapy.
  In terms of efficacy, patients who die before achieving therapeutic success will be counted as a failure, and all patients who receive ≥ 1 dose of protocol chemotherapy will be counted as a failure or success. Only subjects who withdraw or die prior to receiving the first dose of protocol chemotherapy will be considered inevaluable and replaced. The evaluation of tolerability and this phase II design will be performed concurrently, i.e., the first enrollees will be counted for both tolerability and efficacy.
Time Frame: At the end of therapy cycle 2 (approximately 2-3 months)
Measure: Number; unit: proportion
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 2
proportion | 0

3. Secondary Outcome: 3-year Event Free Survival (EFS)
Description: We will use the Kaplan-Meier method to describe event-free survival. EFS will be defined as the time from enrollment to death, relapse, or refractory disease with event-free subjects' time censored at the date of last follow-up.
Time Frame: 3 years after enrollment of the last participant
Measure: Number; unit: Percentage of participants
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 2
Percentage of participants | 0

4. Secondary Outcome: 3-year Overall Survival (OS)
Description: We will use the Kaplan-Meier method to describe overall survival. Overall survival will be defined as the time from enrollment to death, with living subjects' time censored at the date of last follow-up
Time Frame: 3 years after enrollment of the last participant
Measure: Number; unit: Percentage of participants
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 2
Percentage of participants | 0

5. Secondary Outcome: Median Time to Neutrophil Recovery
Description: The time to neutrophil recovery will be summarized using descriptive statistics. If there are no deaths prior to recovery of neutrophils, nonparametric confidence intervals for the median time to recovery will be computed by inverting the sign test. Otherwise, we will compute cumulative incidence curves to describe the time to platelet and neutrophil recovery while adjusting for competing events.
Time Frame: From start of therapy to completion of therapy (approximately 1 year)
Measure: Median (Full Range); unit: Days
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 2
Days | 14.5 [12 to 17]

6. Secondary Outcome: Time to Platelet Recovery
Description: The time to platelet recovery will be summarized using descriptive statistics. If there are no deaths prior to recovery of platelets, nonparametric confidence intervals for the median time to recovery will be computed by inverting the sign test. Otherwise, we will compute cumulative incidence curves to describe the time to platelet and neutrophil recovery while adjusting for competing events.
  Due to the small number of patients enrolled, the data is presented by patient.
Time Frame: From start of therapy to completion of therapy (approximately 1 year)
Population: Platelet recovery for Patient #1 could not be determined due to transfusions.
Measure: Number; unit: days
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 1
days | 15

7. Secondary Outcome: 1-year Cumulative Incidence of Acute Graft Versus Host Disease (GVHD)
Description: Children's Oncology Group (COG) Stem Cell Committee Consensus Guidelines for Establishing Organ Stage and Overall Grade of Acute Graft Versus Host Disease (GVHD) were used. Overall clinical grade was based on the highest stage obtained:
  * Grade 0: no stage 1-4 of any organ
  * Grade I: stage 1-2 skin and no liver or gut involvement
  * Grade II: stage 3 skin, or stage 1 liver involvement, or stage 1 GI
  * Grade III: stage 0-3 skin, with stage 2-3 liver, or stage 2-3 GI
  * Grade IV: stage 4 skin, liver or GI involvement
Time Frame: From start of therapy through completion of therapy (approximately 1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 2
Participants
  Stage 0 | 0
  Stage I | 0
  Stage II | 0
  Stage III | 2
  Stage IV | 0

8. Other Pre Specified Outcome: Percent Donor Chimerism
Description: Percent donor chimerism in blood and bone marrow.
Time Frame: At weeks 1, 2, 3, and 4 after infusion of HPC-A
Measure: Mean (Full Range); unit: Percentage of donor chimerism
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 2
Percentage of donor chimerism
  Week 1 | 79.5 [61 to 98]
  Week 2 | 99 [98.5 to 99.5]
  Week 3 | 99.5 [99.8 to 99.5]
  Week 4 | 100 [100 to 100]

9. Secondary Outcome: 1-year Cumulative Incidence of Chronic Graft Versus Host Disease (GVHD)
Description: All grades of GVHD will be reported.
Time Frame: From start of therapy through completion of therapy (approximately 1 year)
Population: No patient survived long enough to evaluate chronic GVHD.
Arm/Group | Myeloid Malignancies
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date of participant start of therapy until off study date (up to 8 months).
Arm/Group | Myeloid Malignancies
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloid Malignancies (N=2)
Heart failure (Cardiac disorders) | 1 (1)
Genderal disorders and administration site conditions (General disorders) | 1 (1)
Pulmonary hypertention (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloid Malignancies (N=2)
Graft Versus Host Disease (Immune system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (13)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions (General disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (2)
Lung infection (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Splenic infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (5)
Blood bilirubin increased (Investigations) | 2 (2)
GGT increased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 2 (15)
Neutrophil count decreased (Investigations) | 2 (4)
Platelet count decreased (Investigations) | 2 (22)
White blood cell decreased (Investigations) | 2 (7)
Acidosis (Metabolism and nutrition disorders) | 2 (3)
Alkalosis (Metabolism and nutrition disorders) | 2 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (14)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (5)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated in May 2017 due to poor accrual and because of competing protocols.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Initial Protocol (2015-04-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT02433483/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Version 1.0 (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT02433483/Prot_SAP_001.pdf